CLINICAL TRIAL: NCT02795143
Title: Evaluating the Effect of Isotretinoin in Regulatory T-cell Function in Adverse Cutaneous Drug Eruptions (ACDEs): A Pilot Study
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: PI (Responsible Party) transferred to new institution prior to enrollment and protocol was closed.
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2016P000845
Record Dates: First submitted 2016-06-06; First posted 2016-06-09 (Estimated); Last update posted 2023-06-07 (Actual); Status verified 2016-12

CONDITIONS: Toxic Epidermal Necrolysis
Keywords: TEN
MeSH Terms: conditions — Stevens-Johnson Syndrome | interventions — Isotretinoin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Isotretinoin (Experimental): Isotretinoin will be given at the following dosage:
  Dosing will be as listed on the table below.
  Weight in Kg Total Daily Dose 40-49 Kg 40mg 50-89 Kg 80mg 90-150 Kg 120mg
  Interventions: Drug: Isotretinoin
- Placebo (Placebo Comparator): Subjects will be given placebo capsules twice a day.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Isotretinoin
  Arms: Isotretinoin
Other: Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine whether isotretinoin is helpful in treating patients with an adverse cutaneous drug eruption known as toxic epidermal necrolysis (TEN).

DETAILED DESCRIPTION:
Toxic epidermal necrolysis (TEN) is a potentially life-threatening skin disorder characterized by widespread redness, blistering and peeling of skin.

Currently, supportive care in the standard treatment for patients with TEN. Isotretinoin, an FDA-approved medication commonly used for treating severe acne induces differentiation of certain inflammatory cells and thus may potentially be helpful in treating patients with TEN.

This is a randomized, placebo-controlled, double-blind, pilot study comparing the efficacy and safety of isotretinoin versus placebo in treating subjects with toxic epidermal necrolysis (TEN).

Approximately 40 subjects who satisfy all inclusion and exclusion criteria will be randomly assigned in a 1:1 ratio to either isotretinoin or placebo which they will take for up to 14 days. The end of the study is defined as the time the subject is discharged from the hospital. Participants will primarily be assessed for percent body surface affected (BSA) and number of days of hospitalization.

ELIGIBILITY:
Inclusion Criteria:

1. 18 - 69 years of age
2. Has biopsy-proven toxic epidermal necrolysis (TEN)
3. If female, should not be of childbearing potential defined as:

   * Have not had menstrual periods for 12 months in a row (menopause) OR
   * Had bilateral oophorectomy or total hysterectomy OR
   * Have a ovarian disorder that would make pregnancy not possible

Exclusion Criteria:

1. Unknown HIV status and unwilling to undergo HIV testing
2. Women of childbearing potential
3. Pregnancy
4. Breastfeeding
5. Fasting serum triglyceride levels >25% of upper limit of normal
6. Aspartate aminotransferase (AST), alanine aminotransferase (ALT), and alkaline phosphatase levels >2× upper limit of normal (ULN)
7. Known allergy to isotretinoin
8. History of suicidal attempt, psychosis, major depression or other serious mood disorders
9. Currently taking vitamin A supplements, tetracyclines, phenytoin, corticosteroids, IVIg or St. John's Wort
10. Has any condition that, in the opinion of the investigator, would make participation not be in the best interest (for example, compromise the well-being) of the participant or that could prevent, limit, or confound the protocol-specified assessments
11. Participation in an interventional study within the past 30 days.

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-11; Primary Completion 2020-06 (Estimated); Study Completion 2020-06 (Estimated)

PRIMARY OUTCOMES:
Number of days of hospitalization | up to 14 days
  Number of days patient will be hospitalized.

SECONDARY OUTCOMES:
Percent of body surface affected (BSA) | up to 14 days
  Maximum body surface affected with TEN.

CONTACTS AND LOCATIONS:
Overall Officials: Arturo Saavedra, MD, PhD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No